CLINICAL TRIAL: NCT06976060
Title: High-Intensity Interval Training in a Community Gym
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2005507
Record Dates: First submitted 2025-05-09; First posted 2025-05-16 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-05

CONDITIONS: Age-related Strength Loss
Keywords: high-intensity interval training; older adults
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High-Intensity Interval Training (Experimental)
  Interventions: Behavioral: High-Intensity Interval Training

INTERVENTIONS:
Behavioral: High-Intensity Interval Training — High-intensity interval training (HIIT) sessions will occur twice per week, on non-consecutive days. Each training session will last 45-60 minutes and consist of eight functional movement exercises incorporating the entire body (upper body, lower body, core/stability, cycling, and agility). Participants will complete two rounds of the 8-exercise circuit with 2-minutes of rest between rounds. The load/resistance used for each exercise will be self-selected by the participants that equates to 15-18 on the RPE scale. During each round, participants will have 1 minute to complete as many repetitions as possible of a given exercise and then have 1 minute of rest before completing the next exercise - giving the participants a 1:1 exercise-to-rest ratio.

SUMMARY:
This study will deliver a 9 week high intensity interval training (HIIT) class using functional movements within a community based gym. The class will be twice a week. Outcomes are focused on cardiovascular endurance, balance, strength and muscle size and muscle quality changes. The outcomes will be assessed weekly.

DETAILED DESCRIPTION:
We will measure cardiovascular endurance (2-minute Step Test; 2MST), balance (Functional Gait Assessment; FGA), muscular strength (Grip Strength and 5 times sit-to-stand; 5xSTS) and muscle size (thickness) and quality (echo intensity) on a weekly basis over the 9 week HIIT class.

ELIGIBILITY:
Inclusion Criteria:

* no contraindications to exercise (PAR-Q+)
* do not have severe mental impairment (>14 on the SAGE)
* ability to walk 100 ft without the use of an assistive device

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2025-06-03 (Actual); Primary Completion 2025-08-07 (Actual); Study Completion 2025-08-07 (Actual)

PRIMARY OUTCOMES:
2-minute Step Test Performance | Baseline and weekly over the 9 week intervention
  Cardiovascular endurance metric, number of repetitions a single leg is able to complete in 2 minutes.

SECONDARY OUTCOMES:
Functional Gait Asssessment | Baseline and weekly over the 9 week intervention
  Balance metric, reporting the score out of 30 points
5 times sit to stand | Baseline and weekly over the 9 week intervention
  Lower extremity muscular strength. Recording the amount of time to complete 5 sit to stand repetitions.
Grip Strength | Baseline and weekly over the 9 week intervention
  Upper Extremity Strength assessment. Peak grip strength measured with hand held dynamometer.
Muscle Thickness | Baseline and weekly over the 9 week intervention
  Muscle thickness will be recorded via ultrasound
Muscle Echo Intensity | Baseline and weekly over the 9 week intervention
  Ultrasound images of the vastus lateralis will be obtained and echo intensity for the muscle will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- UNMC Engage Wellness Medical Fitness Center, Omaha, Nebraska, United States